CLINICAL TRIAL: NCT06806566
Title: Clinical Evaluation of Carvacrol Loaded Absorbable Gelatin Sponge As a Palatal Bandage After Free Gingival Graft Harvesting : a Randomized Clinical Trial
Brief Title: Assessment of a Carvacrol-loaded Absorbable Gelatin Sponge Used As a Palatal Dressing Following Free Gingival Graft Harvesting: a Randomized Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Amin, Principal Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-011
Record Dates: First submitted 2025-02-03; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Palatal Wound
MeSH Terms: interventions — carvacrol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Biostatistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Absorbable gelatin sponge soaked in carvacrol oil
  Interventions: Other: Carvacrol
- Control Group (Active Comparator): Gelatin Sponge
  Interventions: Other: Gelatin Sponge Sheet

INTERVENTIONS:
Other: Carvacrol — 1-absorbable gelatine sponge soaked in carvacrol oil placed in the palatal donor site.
  Procedure:
  The palatal sites will be anaesthetized with 0.3 ml of a solution of 4% Articaine and 0.001% Adrenalin. Graft harvesting will be performed by basic surgical techniques previously described by Miller (1982). A rectangular shaped piece of mucosa will be harvested from the area of the hard palate by a split-thickness dissection.
  The graft will then be used as it on the recipient bed. The graft dimensions will be recorded (width and length). Denuded palatal area will then be protected using a carvacrol loaded absorbable gelatin sponge (test group)
  Arms: Test Group
Other: Gelatin Sponge Sheet — Absorbable gelatin sponge placed in the palatal donor site
  Procedure:
  The palatal sites will be anaesthetized with 0.3 ml of a solution of 4% Articaine and 0.001% Adrenalin. Graft harvesting will be performed by basic surgical techniques previously described by Miller (1982). A rectangular shaped piece of mucosa will be harvested from the area of the hard palate by a split-thickness dissection.
  The graft will then be used as it on the recipient bed. The graft dimensions will be recorded (width and length). Denuded palatal area will then be protected using a absorbable gelatin sponge(control group).
  Arms: Control Group

SUMMARY:
To evaluate the effect of carvacrol loaded to absorbable gelatin sponge as a palatal bandage on the palatal donor site in post-operative pain reduction after free gingival graft harvesting

ELIGIBILITY:
Inclusion Criteria:

1 - Patients with mucogingival defects scheduled for free gingival graft. 2- Medically free patients 3- Palate with sufficient connective tissue to accommodate soft tissue defects. 4- Good oral hygiene

Exclusion Criteria:

1 - Smokers 2- Pregnancy 3- Medically compromised patients 4- Severe gag reflex 5- Patients allergic to the used agent 6- Occlusal trauma at the site of graft

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Pain | 2 weeks
  Pain score reported by the patient directly through Visual Analogue Scale score (between 0 and 10. 0: no pain, 1: minimal pain, 5:moderate pain, 10: severe pain)

SECONDARY OUTCOMES:
Color Match | 42 days
  On day 3, day 7, day 14, day 21 and day 42, the color of the palatal mucosa will be assessed by comparing it with that of the adjacent and opposite side by using the objective VAS (VAS score 0-10) represented by a continuous line, by a clinician blinded to the treatment group assignment.
  A score of 0 indicates no color match, and a score of 10 indicates excellent color match with the adjacent tissues
Wound Size | 21 days
  To be recorded using (UNC15) periodontal probe to the nearest measurement of 0.5 mm at surgery day, day 3, day 7, day 14 and day 21
Post-Operative Pain (Indirectly) | 3 Weeks
  Postoperative pain, number of analgesic pills taken, and number of days pills were taken were assessed using questionnaires administered at the 3-day and 3-week postoperative appointments.

CONTACTS AND LOCATIONS:
Locations (1):
- The british university in egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided